CLINICAL TRIAL: NCT03815760
Title: Can Blood Flow Restriction Therapy Improve Strength for Shoulder External Rotators Better Than Exercise Alone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Jason Brumitt, Assistant Professor of Physical Therapy, George Fox University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2181055
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Muscular Weakness
Keywords: infraspinatus, external rotators, blood flow restriction
MeSH Terms: conditions — Muscle Weakness | interventions — Blood Flow Restriction Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Exercise with Blood Flow Restriction (Experimental): Subjects will perform the sidelying external rotation exercise 2x a week for 8 weeks.
  The BFR cuff will be applied to the upper arm. Arterial occlusion will be set to 50%.
  Subjects will perform 4 sets (30, 15, 15, 15 reps) with a 30 sec rest period between reps. The occlusion will be maintained for the 8 min treatment period.
  Interventions: Device: Blood Flow Restriction
- Exercise without Blood Flow Restriction (Active Comparator): Subjects will perform the sidelying external rotation exercise 2x a week for 8 weeks.
  This group will not have BFR applied. Subjects will perform 4 sets (30, 15, 15, 15 reps) with a 30 sec rest period between reps.
  Interventions: Device: Blood Flow Restriction

INTERVENTIONS:
Device: Blood Flow Restriction — Subjects will perform sidelying external rotation exercise
  Other Names: Exercise

SUMMARY:
The purpose of this study is to evaluate the ability of blood flow restriction therapy to improve strength of shoulder muscles during the sidelying external rotation (ER) exercise versus a control group who only performs the sidelying ER exercise.

DETAILED DESCRIPTION:
The purpose of this study is to determine if blood flow restriction (BFR) therapy is superior at increasing strength of the shoulder (supraspinatus, infraspinatus, posterior deltoid, and middle deltoid) and increasing tendon size of the supraspinatus and infraspinatus (as determined by diagnostic ultrasound) while performing the sidelying external rotation exercise compared to those who only perform the sideyling external rotation exercise without BFR.

Subjects will be randomized to one of two treatment groups: exercise with BFR or exercise alone. Recruitment will be a sample of convenience consisting of healthy adults (age range 22 to 45). Subjects will perform the sidelying external rotation exercise 2 times a week for an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult (age 18 and older) with no current shoulder pathology

Exclusion Criteria:

1. Current neck, shoulder (or general upper extremity), and/or thoracic spine pathology
2. Shoulder surgery (or general upper extremity surgery) during the prior 6-month time period
3. Cervical/thoracic spine surgery during the prior 1 year
4. Subject having one or more contraindications for BFR training.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Muscular Strength as Measured by Dynamometry | Change from Baseline to 8-weeks
  Use a hand held dynamometer (MicroFet 2) to measure strength of the middle and posterior deltoid, the supraspinatus, and the infraspinatus
Tendon Size as Measured by Diagnostic Ultrasound | Change from Baseline to 8-weeks
  Ultrasound images are capture at pre- and post-test sessions

CONTACTS AND LOCATIONS:
Overall Officials: Jason Brumitt, PhD, Principal Investigator — George Fox University
Locations (1):
- George Fox University School of Physical Therapy, Newberg, Oregon, United States

IPD SHARING:
Plan to Share IPD: No